CLINICAL TRIAL: NCT05101317
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of HMI-115 in Women With Moderate to Severe Endometriosis-Associated Pain Over a 12-Week Treatment Period
Brief Title: A Study to Assess the Efficacy and Safety of HMI-115 in Subjects With Endometriosis-Associated Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Medicine (Nanjing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMI-115EM201
Record Dates: First submitted 2021-10-09; First posted 2021-11-01 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HMI-115 60mg (Experimental): Once Every 2 weeks, subcutaneously injection
  Interventions: Drug: HMI-115
- HMI-115 120mg (Experimental): Once Every 2 weeks, subcutaneously injection
  Interventions: Drug: HMI-115
- HMI-115 240mg (Experimental): Once Every 2 weeks, subcutaneously injection
  Interventions: Drug: HMI-115
- Placebo (Placebo Comparator): Once Every 2 weeks, subcutaneously injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMI-115 — HMI-115 is human monoclonal antibody
  Arms: HMI-115 120mg; HMI-115 240mg; HMI-115 60mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of HMI-115 compared to placebo over a 12 weeks period on subjects with moderate to severe endometriosis-associated pain.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and efficacy of HMI-115 versus a placebo in pre-menopausal women with moderate to severe Endometriosis associated pain.

The study will determine the safety and efficacy of HMI 115 at 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal female subjects, between 18 and 49 years of age, inclusive, at the time of signing informed consent.
2. Subject must have a clinical diagnosis of endometriosis (laparoscopy or laparotomy) as documented by medical records within 10 years before screening.
3. Subject must have a Composite Pelvic Signs and Symptoms Score total score of ≥ 6 with a score of at least 2 for DYS and at least 2 for NMPP at screening.
4. Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

1. Subject is pregnant or breastfeeding or is planning a pregnancy during the study period.
2. Subject has chronic pelvic pain that is not caused by endometriosis or has any other chronic pain syndrome or other chronic therapy, or that would interfere with the assessment of endometriosis-related pain
3. Subject has clinically significant gynecologic condition other than endometriosis
4. Subject has previous history of a severe, life-threatening or other significant sensitivity to any opioids or non-steroidal anti inflammatory drugs (NSAIDS) or any contraindication to their use such as gastrointestinal ulcer or bleeding
5. Subject has history of hysterectomy and/or bilateral oophorectomy
6. Subjects with past or present pituitary tumor growth
7. Subjects has a history of osteoporosis or other metabolic bone disease

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Physicians' Research Options, LLC- Corner Canyon Clinic, Draper, Utah
  - Tidewater Clinical Research/TPW, Norfolk, Virginia
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China
- Poland (2):
  - Instytut Matki i Dziecka, Warsaw, Masovian Voivodeship
  - Specjalistyczna Poradnia Ginekologiczna Gabinet Ginekologiczny Dr med. Janusza Tomaszewskiego, Bialystok, Podlaskie Voivodeship

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in China, the United States of America (USA), and Poland.Total of 310 subjects were screened, of which 142 subjects were randomized. Among them, 36 subjects received HMI-115 60 mg, 36 received HMI-115 120 mg, 35 received HMI-115 240 mg, and 35 subjects were randomized to receive placebo. In the protocol version 5.0, part 2 of the study was deleted and not executed. So no subject was recruited in the former planned part 2 study.
Pre-assignment Details: 1. Screening Period: up to 75 days prior to first dose
  * Screening Visit 1
  * Screening Visit 2 (at least 35 days before Visit 3 to ensure at least 5 weeks Baseline pain score obtained before randomization)
Period: Week1-13
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Started | 36 | 36 | 35 | 35
Completed | 36 | 33 | 35 | 34
Not Completed | 0 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Early Withdrawl | 0 | 0 | 0 | 1
Period: Week 13-25
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Started | 36 | 33 | 35 | 34
Completed | 35 | 30 | 33 | 34
Not Completed | 1 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Patient decide to have oral contraception/refuse to come back | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: PAS：All subjects in the FAS(All randomized subjects who take at least one dose of IMP) who have surgical diagnosis.
Groups:
- Total: Total of all reporting groups
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 24 | 30 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (4.43) | 36.4 (4.99) | 37.4 (5.31) | 38.1 (5.17) | 38.0 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 24 | 30 | 108
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 26 | 27 | 24 | 29 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 13 | 9 | 15 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 15 | 14 | 14 | 15 | 58
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 2 | 5
  China | 12 | 13 | 9 | 15 | 49
  Poland | 14 | 13 | 14 | 13 | 54
Endometriosis duration [Mean (Standard Deviation); unit: months] | 67.2 (37.8) | 57.0 (31.8) | 67.4 (28.7) | 73.7 (27.2) | 66.5 (31.7)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.57 (4.011) | 23.17 (3.220) | 24.40 (4.046) | 23.25 (4.223) | 23.57 (3.873)
DYS NRS [Mean (Standard Deviation); unit: units on a scale] | 6.288 (1.4261) | 6.393 (2.1123) | 5.910 (1.8236) | 5.696 (2.0005) | 6.127 (1.7909)
NMPP NRS [Mean (Standard Deviation); unit: units on a scale] | 3.662 (1.8258) | 3.985 (1.6538) | 4.052 (2.0056) | 3.643 (1.8806) | 3.824 (1.8253)
NSAIDs [Mean (Standard Deviation); unit: pills] | 1.283 (1.2805) | 1.481 (1.7239) | 1.411 (1.4096) | 1.112 (1.1415) | 1.307 (1.3654)
Average Menstrual Bleeding Score [Mean (Standard Deviation); unit: units on a scale] | 2.594 (0.5639) | 2.710 (0.7107) | 2.722 (0.5610) | 2.514 (0.5826) | 2.629 (0.6060)
Monthly Mean Endometriosis Daily Impact Pain Scale [Mean (Standard Deviation); unit: units on a scale]
  DYS | 2.303 (0.4370) | 2.281 (0.6385) | 2.193 (0.5580) | 2.122 (0.6031) | 2.223 (0.5626)
  NMPP | 1.390 (0.6000) | 1.529 (0.5878) | 1.588 (0.6516) | 1.435 (0.6191) | 1.481 (0.6102)
  DYSP | 0.906 (0.6429) | 1.158 (0.9168) | 1.102 (0.8189) | 1.358 (0.6214) | 1.149 (0.7483)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dysmenorrhea (DYS) Measured by Numeric Rating Scale (NRS) From Baseline to Week 12 (Percentage Change)
Description: The Numeric Rating Scale for dysmenorrhea ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Time Frame: Baseline, Week 12
Population: PAS: All randomized subjects with at least 1 dose with surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
percentage of change from baseline | -27.35 (9.568) | -34.72 (9.630) | -41.57 (10.234) | -18.61 (8.859)

2. Primary Outcome: Change in Dysmenorrhea (DYS) Measured by Numeric Rating Scale (NRS) From Baseline to Week 12（Absolute Score Change）
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: All randomized subjects with at least 1 dose with surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
score on a scale | -2.57 (0.542) | -3.29 (0.546) | -3.26 (0.579) | -2.31 (0.502)

3. Secondary Outcome: Change in Dysmenorrhea (DYS) Measured by Numeric Rating Scale(NRS) From Baseline to Week 24 (Percentage Change)
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: PAS: All randomized subjects who had at least 1 dose with surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
percentage of change from baseline | -6.86 (11.912) | -21.82 (12.039) | -14.07 (12.736) | 3.97 (10.898)

4. Secondary Outcome: Change in Non-menstrual Pelvic Pain (NMPP) Measured by Numeric Rating Scale (NRS) From Baseline to Week 12 and 24 (Percentage Change)
Description: The Numeric Rating Scale for non-menstrual pelvic pain (NMPP) ranges 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Time Frame: Baseline, week 12 and 24
Population: PAS: All randomized subjects with at least 1 dose with Surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
percentage of change from baseline
  Week12 %CFB | -33.74 (10.283) | -47.48 (10.363) | -51.66 (11.157) | -27.61 (9.577)
  Week24 %CFB | -11.22 (15.063) | -56.62 (15.252) | -38.05 (16.341) | -33.30 (13.800)

5. Secondary Outcome: Change in Dyspareunia (DYSP) Measured by NRS From Baseline to Week 12 and 24 (Percentage Change)
Description: The Numering Rating Score for dyspareunia ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Time Frame: Baseline, week 12 and 24
Population: All randomized subjects with at least 1 dose with surgical diagnosis and responsed having sexual intercourse at both baseline and endpoints
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 17 | 15 | 18 | 22
percentage of change from baseline
  Week12 %CFB | -7.01 (19.073) | -38.43 (20.420) | -11.70 (22.342) | -24.98 (16.627)
  Week24 %CFB | -2.32 (28.065) | -61.91 (30.048) | 3.47 (30.259) | -13.17 (22.422)

6. Secondary Outcome: Change From Baseline (CFB) in the Monthly Mean Endometriosis Daily Impact Pain Scale for DYS, NMPP and DYSP
Description: Endometriosis Daily Impact Pain Scale ranges from 0 (none) to 3 (severe) as recorded in a daily electronic diary. The higher scores mean worse outcome.
Time Frame: Baseline, week 12 and 24
Population: All randomized subjects with at least 1 dose with surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
score on a scale
  Week 12 DYS | -0.83 (0.184) | -1.06 (0.185) | -1.13 (0.197) | -0.79 (0.172)
  Week 24 DYS | -0.60 (0.192) | -0.87 (0.194) | -0.66 (0.205) | -0.48 (0.176)
  Week12 NMPP | -0.49 (0.119) | -0.61 (0.119) | -0.69 (0.128) | -0.46 (0.110)
  Week24 NMPP | -0.42 (0.162) | -0.78 (0.165) | -0.63 (0.178) | -0.49 (0.149)
  Week12 DYSP | -0.01 (0.169) | -0.48 (0.173) | -0.16 (0.187) | -0.02 (0.149)
  Week24 DYSP | -0.19 (0.210) | -0.69 (0.230) | -0.28 (0.222) | -0.13 (0.179)

7. Secondary Outcome: Change From Baseline (CFB) by Visit in Permitted Rescue Medication Use
Description: Assessment was based on average pill counts at each apecific period od days
Time Frame: Baseline, week 12 and 24
Population: PAS: All randomized subjects with at least 1 dose with surgical diagnosis
Measure: Mean (Standard Deviation); unit: pill
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
pill
  CFB Week12 Average pill count Tier 1 | -0.656 (1.4020) | -0.463 (0.9113) | -1.001 (1.4900) | -0.384 (0.8579)
  CFB Week24 Average pill count Tier1 | -0.394 (1.4724) | -0.643 (1.8192) | -0.590 (1.1144) | -0.414 (0.9968)

8. Secondary Outcome: Change in Menstrual Period Heaviness (Bleeding) From Baseline by Visit
Description: Assessment was based on tampons or pads used. 0 means no bleeding, 4 means heavy bleeding. Higher score means more bleeding.
Time Frame: Baseline, week 12 and 24
Population: PAS:All ranomized subjects with at least 1 dose with surgical diagnosis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
score on a scale
  CFB Week 12 Average Score | -0.415 (0.7062) | -0.571 (0.6114) | -0.363 (0.6437) | -0.197 (0.4525)
  CFB Week 24 Average score | -0.119 (0.6463) | -0.390 (0.8419) | -0.585 (0.6965) | -0.114 (0.4920)

9. Secondary Outcome: Change in Dysmenorrhea(DYS) Measured by Numeric Rating Scale (NRS) From Baseline to Week 24 (Absolute Score Change)
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: PAS: All randomized subjects with at least 1 dose with surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
score on a scale | -1.87 (0.579) | -2.95 (0.585) | -2.18 (0.617) | -1.45 (0.529)

10. Secondary Outcome: Change in Non-menstrual Pelvic Pain (NMPP) Measured by Numeric Rating Scale (NRS) From Baseline to Week 12 and 24 (Absolute Score Change)
Description: The Numeric Rating Scale (NRS) for non-menstrual pelvic pain (NMPP) ranges 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Time Frame: Baseline, Week12, Week24
Population: PAS: All randomized subjects with at least 1 dose with Surgical diagnosis
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 27 | 27 | 24 | 30
score on a scale
  Week12 | -1.46 (0.344) | -1.64 (0.347) | -1.92 (0.373) | -1.36 (0.321)
  Week24 | -1.21 (0.452) | -2.07 (0.457) | -1.67 (0.490) | -1.26 (0.415)

11. Secondary Outcome: Change in Dyspareunia (DYSP) Measured by Numering Rating Score(NRS) From Baseline to Week 12 and 24 (Absolute Score Change)
Description: The Numering Rating Score(NRS) for dyspareunia(DYSP) ranges from 0 (no pain) to 10 (severe pain). Higher scores mean a worse outcome.
Time Frame: Baseline, Week12, Week24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
Number analyzed (Participants) | 17 | 15 | 18 | 22
score on a scale
  Week12 | -0.23 (0.487) | -1.33 (0.489) | -0.90 (0.518) | -0.54 (0.423)
  Week 24 | -1.03 (0.547) | -2.13 (0.591) | -1.57 (0.546) | -0.68 (0.456)

ADVERSE EVENTS:
Time Frame: All AEs and SAEs will be collected from the signing of informed consent form until the end of study participation （About 34 weeks）
Arm/Group | HMI-115 60mg | HMI-115 120mg | HMI-115 240mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 1/24 | 0/30
Other Adverse Events (participants affected / at risk) | 15/27 | 16/27 | 18/24 | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMI-115 60mg (N=27) | HMI-115 120mg (N=27) | HMI-115 240mg (N=24) | Placebo (N=30)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HMI-115 60mg (N=27) | HMI-115 120mg (N=27) | HMI-115 240mg (N=24) | Placebo (N=30)
Injection site pruritus (General disorders) | 1 (5) | 2 (5) | 3 (12) | 1 (2)
Injection site rash (General disorders) | 2 (2) | 3 (5) | 1 (4) | 0 (0)
Injection site reaction (General disorders) | 1 (5) | 2 (4) | 2 (9) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 2 (2) | 1 (1)
Vaginal infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 3 months from the time submitted to the sponsor for review. If no response from the sponsor in 3 months, it will be treated as the sponsor agrees the publication.

DOCUMENTS (2):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT05101317/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT05101317/SAP_001.pdf